CLINICAL TRIAL: NCT01603121
Title: A Safety, Tolerability and Bioavailability Study of Lisofylline After Continuous Subcutaneous (12 mg/kg) and Intravenous (9 mg/kg) Administration in Subjects With Type 1 Diabetes Mellitus
Brief Title: Lisofylline as Continuous Subcutaneous and Intravenous Administration in Subjects With Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to enroll sufficient number of subjects
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, David C. Lieb, MD, Dr., Eastern Virginia Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DL-001
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: lisofylline
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — lisofylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lisofylline subcutaneous (Experimental): Lisofylline 12mg/kg as a continuous subcutaneous infusion over a 10 hours period
  Interventions: Drug: Lisofylline
- Lisofylline intravenous (Experimental): Lisofylline 9 mg/kg as a continuous intravenous infusion over a 10 hours period
  Interventions: Drug: Lisofylline

INTERVENTIONS:
Drug: Lisofylline — Lisofylline single dose of 9 mg/kg continuous intravenous infusion over a 10 hour period, and lisofylline single dose of 12 mg/kg continuous subcutaneous infusion over a 10 hour period during the alternate period 1 week apart.

SUMMARY:
The primary goal of the study is to investigate the safety and tolerability of the investigational drug lisofylline, when administered under the skin or in the vein, in people with type 1 diabetes. A second aim is to determine how much drug is available in the blood after injection under the skin, compared to injection in the vein.

DETAILED DESCRIPTION:
This is an open-label, randomized, crossover study in subjects with type 1 diabetes. There are two treatment periods separated by approximately one week. One treatment will consist of a 10 hour subcutaneous infusion of lisofylline, and the other treatment will consist of a 10 hour intravenous infusion of lisofylline.

Eligible subjects will be admitted to the Infusion Center the morning of dosing (Day 1, Day 7) during each treatment period, receive their assigned dose of study drug on Day 1 and Day 7, and will remain confined to the Infusion Center until approximately 3 hours following the start of study drug administration for the remaining blood draws. The subjects will then be escorted to the Sleep Center of Eastern Virginia Medical School for an overnight stay during which time their heart rate and oxygen saturation will be monitored by pulse oximetry. The next morning the subjects will return to the Infusion Center for a final blood draw and physical examination. The Infusion Center and the Sleep Disorders Center are both within Sentara Norfolk General Hospital.

All subjects will be assigned to a treatment sequence according to a randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults between the ages of 18 and 45 years of age
* Ability to understand and provide written informed consent
* Ability to complete the study in compliance with the protocol
* If female, subjects must be non-pregnant and non-lactating, and willing to use appropriate and adequate contraception during the study
* If male, subjects must be willing to use effective birth control during the study
* Weight at least 50 kgs (110 lbs)
* Body mass index between 18.5 and 30 kg/m2
* QTc < 450 msec at screening
* Clinical diagnosis of type 1 diabetes at least 2 years prior to screening
* Treatment with insulin for at least 1 year and on a stable dose for at least 3 months prior to screening (dose must be < 0.8 units/kg/day)
* Subjects must self-monitor blood glucose levels at least daily
* HbA1c 6-9%
* Serum c-peptide level < 0.6 ng/mL
* Serum creatinine < 1.5 mg/dL for males and < 1.4 mg/dL for females
* Negative hepatitis B, hepatitis C and HIV testing at screening or within 3 months of screening
* Subjects must be free from clinically significant abnormal findings at the time of screening (to include abnormalities on examination, medical history, electrocardiogram, clinical laboratory testing); to be determined by principal investigator

Exclusion Criteria:

* Subjects with significant stomach, liver, kidney or heart disease, including high blood pressure, stroke or other blood vessel disease. Significant eye problems due to diabetes, diabetic nerve disease, or non-healed diabetic foot ulcers
* Personal or family history of long QTc syndrome
* History of clinically significant changes in orthostatic blood pressure
* Clinically significant changes in orthostatic blood pressure at screening
* History of peptic ulcer disease and/or gastrointestinal bleeding/perforation
* History or presence of proliferative retinopathy, severe non-proliferative retinopathy, macular edema or presence of untreated diabetic eye disease
* History of severe peripheral or autonomic neuropathy in the opinion of the study physician
* History of hypoglycemia unawareness, and/or episodes of severe hypoglycemia within 60 days of screening
* Diagnosis of type 2 diabetes, based upon subject report
* Use of oral antihyperglycemic medications, pentoxyifylline, and/or theophylline
* Use of any drug therapy that directly affects gastrointestinal motility
* History of any significant drug allergy
* History of difficulty with phlebotomy
* Use of any recreational drugs within the past year or a previous history of drug or alcohol abuse
* Positive results from a screen for alcohol or substances of abuse at screening or upon admission to the study site
* Current smoker or user of any tobacco products
* Use of prescription medications is acceptable at the Principal Investigator's discretion if they have been part of a stable drug regimen documented for the last 60 days. Drug therapy should be held the morning of Day 1 and Day 7 at the Principal Investigator's discretion
* use of any over-the-counter drugs or herbal preparations within 72 hours prior to receiving study drug
* Consumption of any caffeine-containing foods or beverages within 24 hours prior to receiving study drug
* Consumption of alcohol within 24 hours prior to admission to the study site
* Consumption of any grapefruit or grapefruit-containing juices within 72 hours prior to receiving study drug
* Use of an investigational drug or product, or participation in a drug research study within 30 days prior to receiving drug
* Prior exposure to lisofylline
* Donation of blood (1 pint or more) within 30 days or plasma within 7 days of receiving study drug
* Any condition which in the opinion of the study investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he or she took part in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Lieb, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School Strelitz Diabetes Center, Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisofylline Subcutaneous First, Then Lisofylline Intravenous: Lisofylline 12mg/kg as a continuous subcutaneous infusion over a 10 hours period
  Lisofylline: Lisofylline single dose of 9 mg/kg continuous intravenous infusion over a 10 hour period, and lisofylline single dose of 12 mg/kg continuous subcutaneous infusion over a 10 hour period during the alternate period 1 week apart.
- Lisofylline Intravenous First, Then Lisofylline Subcutaneous: Lisofylline 9 mg/kg as a continuous intravenous infusion over a 10 hours period
  Lisofylline: Lisofylline single dose of 9 mg/kg continuous intravenous infusion over a 10 hour period, and lisofylline single dose of 12 mg/kg continuous subcutaneous infusion over a 10 hour period during the alternate period 1 week apart.
Period: First Intervention, 10 Hours
Arm/Group | Lisofylline Subcutaneous First, Then Lisofylline Intravenous | Lisofylline Intravenous First, Then Lisofylline Subcutaneous
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Second Intervention, 10 Hours
Arm/Group | Lisofylline Subcutaneous First, Then Lisofylline Intravenous | Lisofylline Intravenous First, Then Lisofylline Subcutaneous
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled into the study were included in the baseline analysis.
Groups:
- All Study Participants: Lisofylline: Lisofylline single dose of 9 mg/kg continuous intravenous infusion over a 10 hour period, and lisofylline single dose of 12 mg/kg continuous subcutaneous infusion over a 10 hour period during the alternate period 1 week apart.
Arm/Group | All Study Participants
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Study Drug
Description: Subjects will be monitored for adverse events both during and after the study drug infusion and will undergo physical examinations, electrocardiograms and clinical safety laboratory tests.
  Study staff will contact subjects within 5 days after each dosing period and approximately 30 days after the 2nd dosing period, to review laboratory results and to ask the subject about any changes in health that they have experienced. Should the subject require an in-person evaluation, this will be arranged with the principal or sub-investigator promptly.
Time Frame: 1 month
Arm/Group | Lisofylline Subcutaneous | Lisofylline Intravenous
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Study Drug Bioavailability After Subcutaneous and Intravenous Infusion
Description: Blood will be collected for determination of lisofylline concentrations at various predetermined time points during the infusions, and 10 and 24 hours following infusion completion. This will help to determine if subcutaneous infusion over 10 hours results in similar lisofylline plasma concentrations as with intravenous infusion.
Time Frame: 24 hours
Arm/Group | Lisofylline Subcutaneous | Lisofylline Intravenous
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluation of Early Efficacy of Study Drug
Description: Blood draws will be performed at predetermined time points during and after the infusions in order to measure serum cytokine and chemokine concentrations, as well as to measure plasma STAT 4 and phosphorylated STAT 4 (markers of lisofylline efficacy).
Time Frame: 24 hours
Arm/Group | Lisofylline Subcutaneous | Lisofylline Intravenous
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were assessed for through investigator assessment during the treatment period, and planned phone calls with patient following treatment periods.
Arm/Group | Lisofylline Subcutaneous | Lisofylline Intravenous
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisofylline Subcutaneous (N=1) | Lisofylline Intravenous (N=1)
Syncope (General disorders) | 0 (0) | 1 (1) — Syncope may have been related to lisofylline, though was also taking an ACE-inhibitor, and in retrospect this medication should have been held during the study period. The patient responded immediately to a change in positioning/fluid hydration.
Hypotension (General disorders) | 0 (0) | 1 (1) — Hypotension may have been related to lisofylline, though was also taking an ACE-inhibitor, and in retrospect this medication should have been held during the study period. The patient responded immediately to a change in positioning/fluid hydration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisofylline Subcutaneous (N=1) | Lisofylline Intravenous (N=1)
Dizziness (General disorders) | 1 (1) | 0 (0) — Subject reported a brief period of dizziness one day after subcutaneous infusion of lisofylline.

LIMITATIONS AND CAVEATS:
Early termination due to difficulty recruiting subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No